CLINICAL TRIAL: NCT00362687
Title: GMB: Phase IV, Multicenter, Randomized, Open-Label Pilot Study of Truvada (TDF+FTC) or Emtricitabine (FTC) Alone Versus HAART Interruption in HIV-Infected Patients Who Need to Interrupt HAART and Who Are Infected With HIV Isolates Containing at Least 2 TAMs (or K65R) and M184V
Brief Title: GMB: Study of Truvada (TDF+FTC) or Emtricitabine (FTC) Alone Versus HAART Interruption in HIV-Infected Patients With Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Pedro Ferrer, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-ES-164-0151
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: HIV Infections
Keywords: HIV, HAART
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Truvada 1 tablet once a day.
  Interventions: Drug: Truvada (TDF+FTC) alone; Procedure: No HAART
- 2 (Experimental): Emtricitabine 1 capsule once a day
  Interventions: Drug: FTC alone; Procedure: No HAART

INTERVENTIONS:
Drug: Truvada (TDF+FTC) alone — tenofovir DF 300 mg and emtricitabine 200 mg in a fixed dose tablet formulation
  Arms: 1
Drug: FTC alone — emtricitabine 200 mg
  Arms: 2
Procedure: No HAART — No HAART

SUMMARY:
Many patients who already harbor drug-resistant HIV require interruption of HAART due to poor compliance, poor quality of life, toxicity or development of resistance. In these patients interruption of HAART has a negative impact on patient immune status due to the reemergence of wild-type virus which is in general more pathogenic than HIV isolates containing resistance mutations. There is a need for "bridging" antiretroviral regimens that might prolong time off conventional HAART whilst waiting for a new regimen that is either fully suppressive or less toxic or less demanding for the patient.

DETAILED DESCRIPTION:
Virological failure associated with the appearance of resistant mutations is still common in patients receiving HAART. When HAART fails patients and clinicians can chose from three different courses of action:

1. Switch therapy to a new salvage regimen based on the results of resistance testing.

   Success of the new salvage regimen is maximized if the new regimen includes antiretroviral drugs without cross-resistance with previous failed drugs or, preferably,new classes of drugs. In general, rescue regimens are more complicated for patients due to its higher pill burden; more frequent dosing and sometimes need for parenteral therapy (Enfuvirtide).
2. Stop therapy. This strategy is feasible in patient with relatively preserved immune function. Time off antiretroviral therapy would be highly dependent on previous nadir CD4 cell count (the lowest the nadir, the more rapidly patients loses CD4 cells). In patients with multidrug resistant virus this strategy is used with the goal of achieving virus reversion towards wild-type forms. Reversion towards wild-type virus would theoretically "resensitize" HIV to prior failed drugs. Unfortunately, a number of investigations have suggested that the loss of CD4 cell count occurred during the time off therapy might not be regained after starting rescue therapy. In addition, reversion towards wild type virus does not appear to be associated with a more favourable outcome of rescue therapy.
3. Maintain failing therapy. This strategy has the potential advantage of decreasing the rate of CD4 cell loss. It is known that certain mutations of HIV decrease viral fitness and produce a less pathogenic virus. Consequently, compared to wild-type virus, CD4 destruction is decreased in the presence of resistance mutations. The very important risk inherent to this strategy is the accumulation of new antiretroviral mutations if the regimen is maintained. Due to cross-resistance among antiretroviral drugs, accumulation of new mutations decreases the chances of success of a new salvage regimen.

Choosing among these three different strategies depends on a number of important factors.

1. Availability of antiretroviral drugs active against resistant HIV isolates. Clinicians would be more prone to switch to a new salvage regimen if the new regimen contains a new class of drugs and/or at least three drugs without cross resistance with the antiretroviral included in the failing regimen. This scenario is very likely after first or second regimen failure. However, after third regimen failure the possibilities of including at least three active drugs dramatically decrease. For deep salvage the possibilities of constructing a viable rescue regimen often depends on enrolling the patient in a clinical trial of a new antiretroviral (for example CCR5 inhibitors). Enrolment in the trial very often implies that patients have to wait for an undefined period of time until the trial starts.
2. Willingness of patient to switch to a more complicated regimen. After second regimen failure, rescue therapies involve a higher pill burden, more frequent dosing and, in a substantial number of cases, the need of parenteral therapy with enfuvirtide. In this situation it is possible that the patient prefer not to start the new therapy due to the negative impact of the new regimen in his quality of life.
3. Immune status of the patient. In patients with low CD4 cell count stopping therapy can put the patient at risk of developing an opportunistic disease. In general patients and clinicians are reluctant to stop therapy if the current CD4 cell count is below 200-250 cells/mL.

Apart from the setting of virological failure HAART interruption might be needed in patients with well controlled viral replication (HIV viremia persistently below 50 copies/ mL). Possible reasons for HAART interruption in this scenario are:

1. Toxicity of current regimen.
2. Patient desire (for example travel abroad).
3. Poor quality of life related to treatment issues.
4. Poor adherence to current HAART regimen and an impending risk of developing resistance mutations. When a patient stop HAART due to these reasons, wild-type HIV re-emerges with the consequent loss of CD4 cells. Depending on the immune status of the patient and prior CD4 cell nadir time off therapy might be quite limited.

ELIGIBILITY:
Inclusion Criteria:

HIV-1 infection documented by confirmed positive HIV-1 antibody test and/or positive PCR for HIV-1 RNA.

* Adult patients (over 18 years of age).
* Available genotype (current or historical) showing M184V and (≥ 2 TAMs or K65R).
* CD4 cell count ≥ 350 cells/mL.
* Patient request HAART interruption due to any of the following:

  1. Patient is receiving a suppressive HAART regimen but has problems with adherence,quality of life or toxicity AND there is no alternative simpler, less toxic regimen (typically patients with substantial resistance and good virological control while receiving multiple antiretrovirals).
  2. Due to resistance, patient is receiving a non-suppressive HAART regimen but patient is not willing to change to a new, already available, more complicated optimized salvage regimen (typically 3rd or 4th line of therapy).
* For women of childbearing potential, negative urine pregnancy test at screening visit.
* Agreement to take part in the study and sign the informed consent.

Exclusion Criteria:

Patients receiving a non-registered antiretroviral (ARV) drug.

* Patients who have < 50 HIV-RNA copies/mL while receiving an NNRTI.
* Serum HBsAg positive and patient is receiving an anti-HBV active nucleoside/nucleotide.
* Hypersensitivity to one of the components of the dosage forms of TDF or FTC, or previous history of intolerance to one of these drugs.
* Known history of drug abuse or chronic alcohol consumption that in the clinician opinion contraindicates participation in the study.
* Women who are pregnant or breast feeding or females of childbearing potential who do not use an adequate method of contraception according to the investigator's judgment.
* Current active opportunistic infection or documented infection within the previous 4 weeks.
* Documented active malignant disease (excluding Kaposi sarcoma limited to the skin).
* Renal disease with creatinine clearance < 50 mL/min.
* Concomitant use of nephrotoxic or immuno-suppressive drugs (should be stopped prior to enrollment)
* Receiving on-going therapy with systemic corticosteroids, Interleukin-2 (IL-2) or chemotherapy.
* Patients who are not to be included in the study according to the investigator's criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To compare CD4 cell loses 24 weeks after HAART discontinuation | Through 48 weeks

SECONDARY OUTCOMES:
Proportion of patients with re-initiation of HAART within 24 and 48 weeks | Through 48 weeks
To compare CD4 cell loses 48 weeks after HAART discontinuation | Through 48 weeks
To compare HIV viral loads 4, 24 and 48 weeks after HAART discontinuation:time-weighted average change from baseline through 24 and 48 weeks (DAVG24 and DAVG48) for log10 plasma HIV-1 RNA for patients with plasma HIV-1 RNA >50 copies/mL at baseline | Through 48 weeks
To compare HIV viral loads 4, 24 and 48 weeks after HAART discontinuation: time-weighted average change from 4 weeks through 24 and 48 weeks (DAVG24 and DAVG48) for log10 plasma HIV-1 RNA for patients with <50 copies/mL at baseline | Through 48 weeks
To compare HIV viral loads 4, 24 and 48 weeks after HAART discontinuation: proportion of patients with HIV RNA <400 and <50 copies/mL at 4 weeks for subjects with plasma HIV-1 RNA <50 copies/mL at baseline | Through 48 weeks
To compare HIV viral loads 4, 24 and 48 weeks after HAART discontinuation: compare log10 plasma HIV-1 RNA at week 4 for patients with HIV-RNA < 50 copies/mL at baseline. | Through 48 weeks
To compare development of new mutations in the reverse transcriptase gene 24 and 48 weeks after HAART discontinuation. | Through 48 weeks
Proportion of patients with any adverse event. | Through 48 weeks
Proportion of patients for each adverse event. | Through 48 weeks
Distribution of the intensity if each adverse event (the greatest intensity for each adverse event within a patient will be considered). | Through 48 weeks
Distribution of the relationship between the adverse effect and the study drug (the strongest relation with the study drug for each adverse event within each patient will be considered). | Through 48 weeks
Proportion of patients who discontinue the study prematurely (before week 48)due to adverse events. | Through 48 weeks
Changes in patient's quality of life analyses. | Through 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ferrer, Study Director — Gilead Sciences, S.L.
Locations (1):
- Gilead Sciences, S.L., Madrid, Spain